CLINICAL TRIAL: NCT06678581
Title: A Randomized, Double-Blind, Placebo-Controlled, Single or Multiple Dose Escalation Study to Evaluate the Safety, PK Profile, PD Profile and Food Effects of SAP-001 Tablets in Healthy Chinese Subjects and Gout Patients With Hyperuricemia
Brief Title: SAD,MAD and Food Effect Study of SAP-001 Tablets in Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanton Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanton Pharma Pte. Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SAP-001-103
Record Dates: First submitted 2023-08-24; First posted 2024-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAP-001 (Experimental): Four sequentially ascending dose cohorts are set in SAD study. Three sequentially ascending dose cohorts are set in MAD study.
  Interventions: Drug: SAP-001
- Placebo (Experimental): placebo tablets for oral
  Interventions: Drug: Placebo
- A Randomized, Open-label, two-period crossover FE study (Experimental): 12 subjects are randomized in a 1:1 ratio to sequences A (fasting - fed) and B (fed - fasting).
  Interventions: Drug: SAP-001

INTERVENTIONS:
Drug: SAP-001 — Solid Oral Tablet
  Other Names: SAP-001 tablet
  Arms: A Randomized, Open-label, two-period crossover FE study; SAP-001
Drug: Placebo — Solid Oral Tablet
  Other Names: placebo tablet
  Arms: Placebo

SUMMARY:
To evaluate the pharmacokinetics (PK) profile of single or multiple oral doses of SAP-001 tablets in healthy Chinese subjects and gout patients with hyperuricemia.

To evaluate the safety and tolerability of single oral doses of SAP-001 tablets in healthy Chinese subjects and multiple oral doses of SAP-001 tablets in gout patients with hyperuricemia. To evaluate the pharmacodynamics (PD) profile of single oral doses of SAP-001 tablets in healthy Chinese subjects and multiple oral doses of SAP-001 tablets in gout patients with hyperuricemia.

To evaluate the pharmacokinetics profile of SAP-001 tablets in healthy Chinese subjects under fasted/fed conditions.

ELIGIBILITY:
For SAD and FE study

Inclusion Criteria:

* Male or female Chinese subjects between the ages of 18 and 55 years (inclusive of the cutoff value, the time of signing the informed consent shall prevail) in good health (as determined by medical history, physical examination, 12-lead ECG [heart rate > 50 bpm, PR interval < 200 ms, and QRS width < 120 ms], vital sign measurements, and normal or no clinically significant abnormalities in clinical laboratory evaluations as assessed by the investigator (or designee) at screening and Day -1);
* Body mass index between 18 and 28 kg/m2 (including the cutoff value) at screening, not less than 50 kg for men and 45 kg for women;
* Serum uric acid (sUA) level ≤ 420 μmol/L (7 mg/dL) during the screening period and no history of gout;
* Males and females of childbearing potential must agree to use at least one medically acceptable form of contraception (see Appendix for specific contraceptive measures) from screening through 3 months after the last dose;
* The subjects fully understand the purpose, nature, method and possible adverse reactions of the trial, voluntarily acts as a subject, and signs the informed consent form;
* Able to complete trial per protocol requirements.

Exclusion Criteria:

* Clinically abnormal diseases or factors, including but not limited to neurological, cardiovascular, hematological, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immunological, skeletal system diseases or other factors, which investigator considered inappropriate for study participation;
* Subjects with a history of gastrointestinal surgery or resection (subjects who have undergone appendectomy and/or herniorrhaphy may be included in the study);
* Clinically significant liver function test abnormalities define as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times of the upper limit of normal (ULN) or total bilirubin (TBIL) > ULN at screening or baseline (D-1); or history of clinically significant acute or chronic hepatitis (including infectious, metabolic, autoimmune, hereditary, ischemic, or other forms), liver cirrhosis, or liver tumor.

  * Significant cardiovascular diseases, including:

    1. Acute decompensated heart failure, including exacerbation of chronic heart failure, manifests as signs and symptoms requiring hospitalization and/or intravenous diuretic therapy [New York Heart Association (NYHA) class III to IV], or hemodynamically significant valvular disease and/or other vascular obstructive lesions within 3 months prior to the screening visit;
    2. Any of the following within 6 months prior to the screening visit:

       * Significant cardiac, cerebral, and/or carotid artery diseases, including but not limited to acute coronary syndrome, myocardial infarction, stroke, and/or transient ischemic attack, or unsatisfactory recovery or unstable control at screening;
       * Major cardiovascular or percutaneous procedures, including cardiac ablation, coronary revascularization, and carotid angioplasty; cardiovascular disease likely to require surgical or percutaneous intervention during participation in the study or within 6 months of the screening visit;
    3. History of clinically significant cardiac arrhythmia, including but not limited to any of the following:

       * Symptomatic bradycardia and/or symptomatic ventricular arrhythmia within 3 months prior to the screening visit;
       * Second- or third-degree atrioventricular block, sick sinus syndrome, left bundle branch block;
       * QTcF > 450 ms for males and > 470 ms for females prior to screening or randomization;
       * History of QT prolongation, long QT syndrome, or torsade de pointes;
* Subjects with a history of malignancy (excluding basal cell carcinoma) within 5 years before screening;
* History of acute infection within 14 days prior to screening;
* History of prescription drug abuse or illicit drug use within 6 months before screening, or drug abuse screening positive at baseline (D-1);
* Consumption of more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 6 months before screening or consumption of alcoholic products 48 hours before dosing, or positive baseline (D-1) alcohol breath test; participation in strenuous exercise 48 hours before dosing;
* Any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines that affect blood uric acid levels within 14 days prior to the first dose;
* Moderate to severe smoker (more than 10 cigarettes per day) within 6 months prior to screening;
* Subjects who have a history of special diet (eg, coffee and other caffeine-containing and alcoholic beverages, tea, grapefruit, etc.) within 14 days before screening;
* Subjects who become diarrhea for drinking milk are excluded from the food effect group.
* Human immunodeficiency virus (HIV) antibody positive or syphilis (TP) antibody positive;
* Women who have positive blood pregnancy (β-HCG) test at screening period or baseline (D-1) or are lactating or plan to have children from before the first dose to 3 months after the end of the trial;
* Receiving any other study drug within 3 months prior to the first dose of study drug, or planning to use the study drug during the study;
* History of blood donation or blood loss of more than 400 mL within 30 days prior to screening;
* Any other conditions that, in the opinion of the investigator, might affect the subject's ability to give informed consent or to follow the protocol, or that the subject's participation in the trial might affect the trial's results or his/her own safety.

For MAD study

Inclusion Criteria:

* Male or female Chinese subjects between 18 and 65 years of age, inclusive of the cutoff values, the time of signing the informed consent shall prevail;
* Body mass index between 19 and 32 kg/m2 (including cutoff values) at screening;
* Serum uric acid (sUA) ≥ 420 μmol/L (7.0 mg/dL) at screening or baseline (D-1);
* Patients met 2015 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for gout at screening and without risk of acute gout attack;
* Subjects do not use any uric acid-lowering drugs within 2 weeks prior to dosing;
* Males and females of childbearing potential must agree to use at least one medically acceptable form of contraception (see Appendix for specific contraceptive measures) from screening through 3 months after the last dose;
* The subject fully understands the purpose, nature, method and possible adverse reactions of the trial, voluntarily acts as a subject, and signs the informed consent form;
* Able to complete trial per protocol requirements.

Exclusion Criteria:

* Clinically abnormal diseases or factors, including but not limited to neurological, cardiovascular, hematological, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immunological, skeletal system diseases or other factors, which investigator considered inappropriate for study participation;
* Patients with a history of gastrointestinal surgery or resection (subjects who have undergone appendectomy and/or herniorrhaphy may be included in the study);
* Clinically significant liver function test abnormalities define as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times of the upper limit of normal (ULN) or total bilirubin (TBIL) > ULN at screening or baseline (D-1); or history of clinically significant acute or chronic hepatitis (including infectious, metabolic, autoimmune, hereditary, ischemic, or other forms), liver cirrhosis, or liver tumor.
* sCr > 132.6 μmol/L (1.5 mg/dL) and/or eGFR ≤ 60 mL/min/1.73 m2 (calculated by CKD-EPI formula) at screening;
* Significant cardiovascular diseases, including:

  1. Acute decompensated heart failure, including exacerbation of chronic heart failure, manifests as signs and symptoms requiring hospitalization and/or intravenous diuretic therapy [New York Heart Association (NYHA) class III to IV], or hemodynamically significant valvular disease and/or other vascular obstructive lesions within 3 months prior to the screening visit;
  2. Any of the following within 6 months prior to the screening visit:

     * Significant cardiac, cerebral, and/or carotid artery diseases, including but not limited to acute coronary syndrome, myocardial infarction, stroke, and/or transient ischemic attack, or unsatisfactory recovery or unstable control at screening;
     * Major cardiovascular or percutaneous procedures, including cardiac ablation, coronary revascularization, and carotid angioplasty; cardiovascular disease likely to require surgical or percutaneous intervention during participation in the study or within 6 months of the screening visit;
  3. History of clinically significant cardiac arrhythmia, including but not limited to any of the following:

     * Symptomatic bradycardia and/or symptomatic ventricular arrhythmia within 3 months prior to the screening visit;
     * Second- or third-degree atrioventricular block, sick sinus syndrome, left bundle branch block;
     * New or untreated atrial fibrillation [Subjects with atrial fibrillation with stable (at least 6 months) asymptomatic heart rate control on appropriate therapy (which may include anticoagulation) are allowed to enroll in this study];
     * QTcF > 450 ms for males and > 470 ms for females prior to screening or randomization;
     * History of QT prolongation, long QT syndrome, or torsade de pointes;
     * History of cardiac transplantation, or subject on cardiac transplant checklist or use of left ventricular assist device;
* History of prescription drug abuse or illicit drug use within 6 months before screening, or drug abuse screening positive at baseline (D-1);
* Consumption of more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 6 months before screening or consumption of alcoholic products 48 hours before dosing, or positive baseline (D-1) alcohol breath test;
* Any prescription drug, over-the-counter drug, any vitamin product, or herbal medicine that had an effect on serum uric acid level within 14 days prior to the first dose; exceptions can be discussed on a case-by-case basis (e.g., long-term stable use of low dose aspirin) after discussion and agreement between the investigator and the Sponsor;
* Participates in strenuous exercise 48 hours before administration;
* Human immunodeficiency virus (HIV) antibody positive or syphilis (TP) antibody positive;
* Women who have positive pregnancy test or are lactating during the screening period or baseline (D-1) or plan to have children from before the first dose to 3 months after the end of the trial;
* Patients who have received any other investigational drugs within 3 months prior to the first dose of study drug or plan to use investigational drugs during the study;
* History of blood donation or blood loss of more than 400 mL within 30 days prior to screening;
* Patients with a history of malignancy (excluding basal cell carcinoma) within 5 years before screening;
* History of acute infection within 14 days prior to screening;
* Any other conditions that, in the opinion of the investigator, might affect the subject's ability to give informed consent or to follow the protocol, or that the subject's participation in the trial might affect the trial's results or his/her own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | 168 hours
  PK parameters
area under the drug concentration-time curve from time 0 to the last measurable concentration sample collection time t (AUC0-t) | 168 hours
  PK parameters
area under the drug concentration-time curve from time 0 to 168 hours (AUC0-168h) | 168 hours
  PK parameters
time to maximum concentration (Tmax) | 168 hours
  PK parameters
elimination half-life (t1/2) | 168 hours
  PK parameters
cumulative urinary excretion from 0 to 168 h (Ae0-168h) | 168 hours
  PK parameters
cumulative urinary excretion rate, renal clearance (CLR168h) | 168 hours
  PK parameters

SECONDARY OUTCOMES:
Serum uric acid area under curve (AUCUA) | 168 hours
  Pharmacodynamic Endpoints
cumulative excretion of uric acid (AeUA) | 168 hours
  Pharmacodynamic Endpoints
renal clearance (CLRUA) | 168 hours
  Pharmacodynamic Endpoints
serum creatinine area under curve (AUCCr) | 168 hours
  Pharmacodynamic Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Study Director — Shanton Pharma Co., Ltd.
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No